CLINICAL TRIAL: NCT05137405
Title: HOW THE IMPACT OF COVID-19 HOME STAY ORDERS IS AFFECTING THE PHYSICAL, MENTAL AND FINANCIAL HEALTH AMONG OBESE PATIENTS?
Brief Title: THE IMPACT OF COVID-19 AMONG OBESE PATIENTS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Giovanna Pavone, Medical Doctor, University of Foggia
Other Study IDs: 2
Record Dates: First submitted 2021-11-15; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Sleeve gastrectomy — An online survey format was administered to all obese patients on the waiting list for bariatric surgery in our Department of Medical and Surgical Sciences to obtain information about the COVID- 19 pandemic's impact on patients with obesity starting March 09, 2020 until May 18, 2020.

SUMMARY:
BACKGROUND: Stay-at-home orders in response to the Coronavirus 2 (SARSCoV-2) have forced abrupt changes to daily routines.

The aim of our study is to evaluate the impact of the Stay-at-home orders on the waiting list for bariatric surgery in our Department of Medical and Surgical during covid-19 pandemic.

MATERIALS AND METHODS: In this observational retrospective study, from the 9th of March to 18th May 2020, the patients of our Department were invited to answer to a 14-questions multiple-choice questionnaire relative to weight changes, working activity, daily exercise, dietary behaviors, and conditions potentially impacting the nutritional choices

ELIGIBILITY:
Inclusion Criteria:

- Alle obese patients on the waiting list for bariatric surgery in our Department of Medical and Surgical during covid-19 pandemic from March to May 2020

Exclusion Criteria:

- Patients underwent bariatric surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: An online survey format was administered to all obese patients on the waiting list for bariatric surgery in our Department of Medical and Surgical Sciences to obtain information about the COVID- 19 pandemic's impact on patients with obesity starting March 09, 2020 until May 18, 2020.
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2020-03-08 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
evaluate the impact of the Lock-down period on the mental and physical health of obese patients on the waiting list for bariatric surgery in our Department of Medical and Surgical Sciences during covid-19 pandemic. | March - May 2020
  we have used a 14-questions multiple-choice questionnaire relative to weight changes, working activity, daily exercise, dietary behaviors, and conditions potentially impacting the nutritional choices

CONTACTS AND LOCATIONS:
Locations (1):
- Nicola Tartaglia, Foggia, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-11-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT05137405/Prot_000.pdf